CLINICAL TRIAL: NCT02132559
Title: Effect of Dehydroepiandrosterone Administration in Patients With Poor Ovarian Response According to the Bologna Criteria
Status: Completed | Type: Observational
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: NSFC30901601
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2013-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- DHEA administration,no treatment: The patients of study group received DHEA 25 mg orally,three times a day before the IVF cycle. Except for IVF, the control group of patients did not receive any pre-treatment.
  Interventions: Drug: DHEA

INTERVENTIONS:
Drug: DHEA
  Other Names: dehydroepiandrosterone

SUMMARY:
Women with low ovarian reserve typically respond less well to the drugs used to stimulate the ovary during IVF treatment and produce fewer eggs and, as a result, are less likely to fall pregnant either naturally or after fertility treatment. The ideal stimulation regimen for poor responders is currently unknown.

Dehydroepiandrosterone (DHEA) has been reported to improve pregnancy chances for poor responders, and is now utilized by approximately one third of all IVF centers world-wide. However, the current clinical evidence for DHEA on improvement of ovarian response and IVF outcome is insufficient. The validity of the results of the former studies, especially the varied inclusion criteria used to specify poor responders, is a subject of debate. Recently a uniform definition on poor ovarian response, the Bologna criteria, has been proposed by the European Society for Human Reproduction and Embryology(ESHRE). However, no studies have been performed study to evaluate the potential effects of DHEA supplementation according to these standards.

The purpose of this study is to assess the impact of DHEA supplementation on IVF outcome of poor ovarian responders that fulfill the Bologna criteria.

ELIGIBILITY:
Inclusion Criteria:

Patients with poor ovarian response according to the Bologna criteria

Exclusion Criteria:

women aged > 45 years or baseline follicle stimulating hormone(FSH)levels >40 IU/l.

Ages: 23 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients were stratified according to the Bologna criteria for poor ovarian response. Poor responders were classified with at least two of the three following criteria: (I) advanced maternal age (≥40 years) or any other risk factor for POR; (II) a previous POR(≤3 oocytes with a conventional ovarian stimulation protocol); and (III) an abnormal ovarian reserve test (ORT): antral follicle count (AFC) < 5-7 or serum anti-Mullerian hormone (AMH) <0.5-1.1 ng/mL, as described by the Bologna criteria
Sampling Method: Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rates | 12 weeks after gestation.

SECONDARY OUTCOMES:
Clinical pregnancy rate | 28 days after the embryo transfer
the number of retrieved oocytes | 36-37 hrs after hCG administration
Fertilization rate | on day 1 after oocyte retrieval
Cleavage rate | on day 2 or 3 after oocyte retrieval
Implantation rate | 28 days after the embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Guijin Zhu, Study Director — Reproductive Medicine Center, Tongji Hospital, Tongji Medicine College, Huazhong University of Science and Technology
Locations (1):
- Reproductive Medicine Center, Tongji Hospital, Tongji Medicine College, Huazhong University of Science and Technology, Wuhan, Hubei, China